CLINICAL TRIAL: NCT07074041
Title: The Role of Radiomic Analysis in Spectral Domain Optical Coherence Tomography Imaging of Acquired Vitelliform Lesions.
Brief Title: Radiomic Analysis in OCT Imaging of Acquired Vitelliform Lesions.
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Gilda Cennamo, MD, Federico II University
Other Study IDs: 05809856 Federico II
Record Dates: First submitted 2025-06-12; First posted 2025-07-20 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: VITELLIFORM LESIONS
Keywords: vitelliform lesion; oct; radiomics
MeSH Terms: conditions — Ornithine Carbamoyltransferase Deficiency Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study group: The study population includes patients diagnosed with acquired vitelliforms lesions (aVLs), defined by hyperautofluorescent material on fundus autofluorescence (FAF) and hyperreflective subretinal material on structural optical coherence tomography (OCT).

SUMMARY:
Vitelliform lesions (VLs) are subretinal accumulations of yellowish material on fundoscopy that correspond to hyperautofluorescent material on fundus autofluorescence (FAF) and hyperreflective subretinal material on structural optical coherence tomography (OCT).

VLs are characterised by dynamic changes with progressive resorption of material and are associated with the appearance of visual symptoms, such as reduced visual acuity. The appearance of symptoms and changes in the characteristics of the VLs on retinal imaging are the basis of a sophisticated differential diagnosis, especially to distinguish a neovascular from a non-vascular sub-type.

To date, additional retinal imaging techniques can be helpful in performing differential diagnosis in unclear cases. Radiomics is a quantitative approach to medical imaging that can extract many features to improve medical diagnosis and assess response to treatment.

The aim of this study is to evaluate the performance of radiomics in the diagnosis of dynamic changes in VLs.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of acquired vitelliform lesions

Exclusion Criteria:

* age < 18 years
* axial length higher than 26 mm
* the presence of clinically significant cataract
* the presence of significant concomitant ocular or systemic diseases (such as diabetic retinopathy, uveitis, glaucoma)
* known retinal disorders that could cause vitelliform lesions or retinal fluid (AMD, neovascularization, tractional pathologies, toxic or paraneoplastic syndromes)
* inherited dystrophies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study group included all patients, over 18 years old, with a diagnosis of aVLs, evaluated from march 2022 to january 2025.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Features analysis of aVLs OCT | Baseline
  extraction and analysis of radiomic features from OCT images to characterize empty optical spaces and distinguish empty space in dynamic changes of aVLs from the presence of fluid in case of aVLs complicated by neovascularisation

CONTACTS AND LOCATIONS:
Locations (1):
- University of Naples, Federico II, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No